CLINICAL TRIAL: NCT01777568
Title: Supplemental Oxygen and Surgical-site Infections: An Alternating Intervention Controlled Trial.
Brief Title: Supplemental Oxygen in Colorectal Surgery: A Quality Improvement Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Andrea Kurz, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12-891
Record Dates: First submitted 2012-12-20; First posted 2013-01-29 (Estimated); Results first posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: 30% Oxygen Concentration During Colorectal Surgery; 80% Oxygen Concentration During Colorectal Surgery
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: The designated operating-room suite alternated between using either 30% oxygen as tolerated or 80% oxygen for periods of 2 weeks. For example, the first period used 30% oxygen, the second 80% oxygen, and so on. The oxygen concentration during the initial period was randomly designated by the study statistician. But, thereafter, oxygen delivery was not randomized on a per-patient or even per-period basis.
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 30% oxygen (Experimental): Inspired oxygen will be maintained at 30%.
  Interventions: Drug: 30% oxygen
- 80% oxygen (Experimental): Inspired oxygen will be maintained at 80%.
  Interventions: Drug: 80% oxygen

INTERVENTIONS:
Drug: 30% oxygen — Inspired oxygen will be maintained at 30%.
  Arms: 30% oxygen
Drug: 80% oxygen — Inspired oxygen will be maintained at 30%.
  Arms: 80% oxygen

SUMMARY:
Our primary objective is to develop a clinical pathway for care of patients having colorectal surgery at the Clinic. In particular, the investigators would like to determine what intraoperative concentration of oxygen is optimal in our patients.

DETAILED DESCRIPTION:
The investigators therefore propose to test the primary hypothesis that supplemental oxygen (80% versus 30%) reduces the risk of a composite of surgical sites infection and potentially oxygen-related wound complications. Secondarily, the investigators will assess the incremental cost benefit of 80% versus 30% oxygen. As a safety measure, enough oxygen will always be given to maintain oxygen saturation (as determined by pulse oximetry) ≥95%.

ELIGIBILITY:
Inclusion Criteria:

* adult colorectal surgical patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5749 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Kurz, MD, Principal Investigator — Cleveand Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cohen B, Ahuja S, Schacham YN, Chelnick D, Mao G, Ali-Sakr Esa W, Maheshwari K, Sessler DI, Turan A. Intraoperative Hyperoxia Does Not Reduce Postoperative Pain: Subanalysis of an Alternating Cohort Trial. Anesth Analg. 2019 Jun;128(6):1160-1166. doi: 10.1213/ANE.0000000000004002. PMID 31094783
- [Derived] Cohen B, Ruetzler K, Kurz A, Leung S, Rivas E, Ezell J, Mao G, Sessler DI, Turan A. Intra-operative high inspired oxygen fraction does not increase the risk of postoperative respiratory complications: Alternating intervention clinical trial. Eur J Anaesthesiol. 2019 May;36(5):320-326. doi: 10.1097/EJA.0000000000000980. PMID 30865003
- [Derived] Kurz A, Kopyeva T, Suliman I, Podolyak A, You J, Lewis B, Vlah C, Khatib R, Keebler A, Reigert R, Seuffert M, Muzie L, Drahuschak S, Gorgun E, Stocchi L, Turan A, Sessler DI. Supplemental oxygen and surgical-site infections: an alternating intervention controlled trial. Br J Anaesth. 2018 Jan;120(1):117-126. doi: 10.1016/j.bja.2017.11.003. Epub 2017 Nov 23. PMID 29397118

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 30% Oxygen | 80% Oxygen
Started | 2853 | 2896
Completed | 2853 | 2896
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 30% Oxygen | 80% Oxygen | Total
Number analyzed (Participants) | 2853 | 2896 | 5749
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (17) | 52 (17) | 52 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1358 | 1387 | 2745
  Male | 1495 | 1509 | 3004
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 2558 | 2627 | 5185
  Africa American | 235 | 207 | 442
  other | 60 | 62 | 122

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Composite Complications
Description: A composite of complications:
  1. surgical sites infection (organ space / deep)
  2. Anastomotic leak
  3. Intra-abdominal abscess
  4. Sepsis
  5. Wound dehiscence
  6. Death
Time Frame: Postoperative 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 30% Oxygen | 80% Oxygen
Number analyzed (Participants) | 2853 | 2896
Participants | 314 | 314
Statistical Analysis 1: Comparison: 30% Oxygen vs 80% Oxygen; Test type: Superiority; p = 0.85, GEE model; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.85 to 1.14] — Relative Risk: 80% (numerator) vs. 30% (denominator)

2. Secondary Outcome: Number of Participants With Superficial SSI (Surgical Site Infection)
Description: superficial SSI (Surgical Site Infection)
Time Frame: Postoperative 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 30% Oxygen | 80% Oxygen
Number analyzed (Participants) | 2853 | 2896
Participants | 183 | 150
Statistical Analysis 1: Comparison: 30% Oxygen vs 80% Oxygen; Test type: Superiority; p = 0.047, Chi-squared; Risk Ratio (RR) = 0.80, 95% CI 2-sided [0.66 to 1.01]

ADVERSE EVENTS:
Time Frame: 30-day postoperatively
Arm/Group | 30% Oxygen | 80% Oxygen
All-Cause Mortality (participants affected / at risk) | 10/2853 | 20/2896
Serious Adverse Events (participants affected / at risk) | 314/2853 | 314/2896
Other Adverse Events (participants affected / at risk) | 183/2853 | 150/2896
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 30% Oxygen (N=2853) | 80% Oxygen (N=2896)
SSI (organ space/deep) (Infections and infestations) | 112 (112) | 118 (118)
Anastomotic leak (Infections and infestations) | 36 (36) | 34 (34)
Intra-abdominal abscess (Infections and infestations) | 143 (143) | 133 (133)
sepsis (Infections and infestations) | 94 (94) | 96 (96)
wound dehiscence (Infections and infestations) | 43 (43) | 43 (43)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 30% Oxygen (N=2853) | 80% Oxygen (N=2896)
uperficial SSI (Infections and infestations) | 183 (183) | 150 (150)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No